CLINICAL TRIAL: NCT04884802
Title: Tight Perioperative Blood Pressure Management to Reduce Serious Cardiovascular, Renal, and Cognitive Complications: The GUARDIAN Trial
Brief Title: The GUARDIAN Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Daniel Sessler, Professor and Vice President for Clinical and Outcomes Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-MS-24-1026
Record Dates: First submitted 2021-04-05; First posted 2021-05-13 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight blood pressure management (Experimental): In patients assigned to tight blood pressure control, angiotensin converting enzyme inhibitors and angiotensin receptor blockers will not be given the morning of surgery. Other chronic antihypertensives will only be given as necessary to treat hypertension. Norepinephrine or phenylephrine infusion will be infused at a rate sufficient to maintain intraoperative MAP ≥ 85 mmHg.
  Interventions: Procedure: Tight blood pressure management
- Routine blood pressure management (Other): ACEIs, ARBs, and/or calcium channel blockers can be given the morning of surgery if deemed appropriate by the attending anesthesiologist. Intraoperative blood pressure will be managed per clinical routine.
  Interventions: Procedure: Routine blood pressure management

INTERVENTIONS:
Procedure: Tight blood pressure management — Norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg.
  Arms: Tight blood pressure management
Procedure: Routine blood pressure management — ACEIs, ARBs, and/or calcium channel blockers can be given the morning of surgery if deemed appropriate by the attending anesthesiologist. Intraoperative blood pressure will be managed per clinical routine.
  Arms: Routine blood pressure management

SUMMARY:
An international randomized trial to test the primary hypothesis that perioperative tight blood pressure management reduces a composite of major perfusion-related complications (myocardial injury, stroke, non-fatal cardiac arrest, Stage 2-3 acute kidney injury, deep or organ-space infection, sepsis, and death) in the 30 days after major non-cardiac surgery.

The treatments will be: 1) norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg (tight pressure management); or, 2) routine intraoperative blood pressure management (routine pressure management).

DETAILED DESCRIPTION:
Qualifying patients will be randomized 1:1, with random-sized blocks, stratified by site. The treatments will be: 1) norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg (tight pressure management); or, 2) routine intraoperative blood pressure management (routine pressure management).

Tight pressure management: In patients assigned to tight pressure management, angiotensin converting enzyme inhibitors and angiotensin receptor blockers will not be given the morning of surgery. Other chronic antihypertensives will only be given as necessary to treat hypertension. General anesthesia will be induced with propofol or etomidate which will be given in repeated small boluses or target-controlled infusion in an effort to keep mean arterial pressure ≥85 mmHg. Simultaneously, the vasopressor infusion will be adjusted with the same goal. Anesthetic dose, fluid administration, and vasopressor administration will be adjusted with the goal of maintaining the individual designated baseline mean arterial pressure. Invasive or non-invasive advanced hemodynamic monitoring is not required, but should be used when practical. Clinicians should use available information to optimize vascular volume, afterload, and inotropy.

Routine pressure management: In patients assigned to routine pressure management, ACEIs, ARBs, and/or calcium channel blockers can be given the morning of surgery if deemed appropriate by the attending anesthesiologist. General anesthesia will be induced and maintained per routine.

In both groups, other aspects of anesthetic management will be at the discretion of the responsible anesthesiologist, including the types and volumes of various fluids. Volatile or intravenous anesthesia is permitted. There will be no limitation on ancillary vasoactive, chronotropic, and inotropic drugs. Clinicians will be free to use advanced hemodynamic monitoring (e.g., pulse-wave analysis, esophageal Doppler, etc.). Blood products will be given per routine. Similarly, postoperative analgesic management will be per routine and clinician preference. Neuraxial and peripheral nerve blocks are permitted, but epidural catheters should not be activated until surgery is nearly finished.

In all cases, good judgement will predominate.

ELIGIBILITY:
Inclusion Criteria:

1. At least 45 years old;
2. Scheduled for major noncardiac surgery expected to last at least 2 hours;
3. Having general anesthesia, neuraxial anesthesia, or the combination;
4. Expected to require at least overnight hospitalization (planned ICU admission is acceptable);
5. Are designated ASA physical status 2-4 (ranging from mild systemic disease through severe systemic disease that is a constant threat to life);
6. Expected to have direct intraoperative blood pressure monitoring with an arterial catheter;
7. Cared for by clinicians willing to follow the GUARDIAN protocol;
8. Subject to at least one of the following risk factors:

   1. Age >65 years;
   2. History of peripheral arterial disease;
   3. History of coronary artery disease;
   4. History of stroke or transient ischemic attack;
   5. Serum creatinine >175 μmol/L (>2.0 mg/dl) within 6 months;
   6. Diabetes requiring medication;
   7. Current smoking or 15 pack-year history of smoking tobacco;
   8. Scheduled for major vascular surgery;
   9. Body mass index ≥35 kg/m2;
   10. Preoperative high-sensitivity troponin T >14 ng/L or troponin I equivalent, defined as ≥15 ng/L (Abbott assay), 19 ng/L (Siemens assay, [Borges, unpublished]), or 25% of the 99% percentile for other assays - all within 6 months;
   11. B-type natriuretic protein (BNP) >80 ng/L or N-terminal B-type natriuretic protein (NTProBNP) >200 ng/L within six months.

Exclusion Criteria:

1. Are scheduled for carotid artery surgery;
2. Are scheduled for intracranial surgery;
3. Are scheduled for partial or complete nephrectomy;
4. Are scheduled for pheochromocytoma surgery;
5. Are scheduled for liver or kidney transplantation;
6. Require preoperative intravenous vasoactive medications;
7. Have a condition that precludes routine or tight blood pressure management such as surgeon request for relative hypotension;
8. Require beach-chair positioning;
9. Have a documented history of dementia;
10. Have language, vision, or hearing impairments that may compromise cognitive assessments;
11. Have contraindications to norepinephrine or phenylephrine per clinician judgement;
12. Have previously participated in the GUARDIAN trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6254 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Composite of Major Perfusion-Related Complications | During the initial 30 days after major non-cardiac surgery
  The primary outcome is a composite of major perfusion-related complications (myocardial injury, stroke, non-fatal cardiac arrest, Stage 2-3 acute kidney injury, deep or organ-space infection, sepsis, and death) in the 30 days after major non-cardiac surgery.

SECONDARY OUTCOMES:
Number of Participants with Postoperative Delirium | Initial 4 postoperative days.
  The Postoperative 3-Minute Diagnostic Interview for the Confusion Assessment Method (3D CAM) will be used twice daily to assess for the presence of delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (20):
- United States (6):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wake Forest University, Wake Forest, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - The University of Texas Health Science Center at Houston, Houston, Texas
- China (9):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - West China University Hospital, Chengdu
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, Hong Kong
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - The Affiliated Lianyungang Hospital of Xuzhou Medical University, Xuzhou
- University of Thessaly, Larissa, Greece
- IRCCS Regina Elena National Cancer Institute, Rome, Italy
- National Defense Medical College, Tokyo, Japan
- Turkey (Türkiye) (2):
  - Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Bakırköy
  - Konya City Hospital, Konya

IPD SHARING:
Plan to Share IPD: Yes
Each center will retain ownership of its own data. Publication of center-specific data will not be allowed until after the Main Trial Report is published, or two years have elapsed since enrollment of the last patient. The Executive Committee welcomes suggestions for sub-studies based on a partial or the full trial dataset. Sub-studies will be allocated based on importance and novelty of the proposals, and priority will be given to high-enrolling centers. However, all multi-center publications will be on a collaborative basis and include appropriate co-authors. The Executive Committee will do its best to be fair and equitable in assigning sub-studies.
  Data will be shared with external parties on a collaborative basis with approval of the Executive Committee and appropriate data-use agreements.